CLINICAL TRIAL: NCT00565851
Title: A Phase III Randomized Controlled Clinical Trial of Carboplatin and Paclitaxel (or Gemcitabine) Alone or in Combination With Bevacizumab (NSC #704865) Followed by Bevacizumab and Secondary Cytoreductive Surgery in Platinum-Sensitive, Recurrent Ovarian, Peritoneal Primary and Fallopian Tube Cancer. NCI-Supplied Agents: Bevacizumab (NSC #704865)
Brief Title: Carboplatin, Paclitaxel and Gemcitabine Hydrochloride With or Without Bevacizumab After Surgery in Treating Patients With Recurrent Ovarian, Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00587; NCI-2009-00587 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-0205; GOG-0213; CDR0000546714; GOG-0213 (Other: NRG Oncology); GOG-0213 (Other: CTEP); U10CA027469 (NIH); U10CA180868 (NIH)
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Clear Cell Adenocarcinoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Mucinous Adenocarcinoma; Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinofibroma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Clear Cell Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Primary Peritoneal Transitional Cell Carcinoma; Primary Peritoneal Undifferentiated Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Undifferentiated Carcinoma
MeSH Terms: conditions — Adenocarcinoma, Clear Cell; Adenocarcinoma, Mucinous; Brenner Tumor; Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Docetaxel; Gemcitabine; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm I (paclitaxel, docetaxel, carboplatin) (Active Comparator): Patients receive paclitaxel IV over 3 hours or docetaxel IV over 1 hour and carboplatin over 30 minutes on day 1. Treatment repeats every 21 days.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm II (paclitaxel, docetaxel, carboplatin, bevacizumab) (Experimental): Patients receive chemotherapy as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm III (gemcitabine hydrochloride, carboplatin) (Experimental): Patients receive gemcitabine hydrochloride IV over 60 minutes on days 1 and 8 and carboplatin as in Arm I.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Arm IV (gemcitabine hydrochloride, bevacizumab, carboplatin) (Experimental): Patients receive gemcitabine hydrochloride IV as in Arm III, bevacizumab IV and carboplatin IV as in Arm II.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm II (paclitaxel, docetaxel, carboplatin, bevacizumab); Arm IV (gemcitabine hydrochloride, bevacizumab, carboplatin)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm I (paclitaxel, docetaxel, carboplatin); Arm II (paclitaxel, docetaxel, carboplatin, bevacizumab)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
  Arms: Arm III (gemcitabine hydrochloride, carboplatin); Arm IV (gemcitabine hydrochloride, bevacizumab, carboplatin)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (paclitaxel, docetaxel, carboplatin); Arm II (paclitaxel, docetaxel, carboplatin, bevacizumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies carboplatin, paclitaxel and gemcitabine hydrochloride when given together with or without bevacizumab after surgery to see how well it works in treating patients with ovarian, epithelial, primary peritoneal, or fallopian tube cancer that has come back. Drugs used in chemotherapy, such as carboplatin, paclitaxel and gemcitabine hydrochloride work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as bevacizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether combination chemotherapy is more effective when given with or without bevacizumab after surgery in treating patients with ovarian, epithelial, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if surgical secondary cytoreduction in addition to adjuvant chemotherapy increases the duration of overall survival in patients with recurrent platinum sensitive epithelial ovarian cancer, peritoneal primary or fallopian tube cancer.

II. To determine if the addition of bevacizumab to the second-line and maintenance phases of treatment increases the duration of overall survival relative to second-line paclitaxel and carboplatin alone in patients with recurrent platinum sensitive epithelial ovarian cancer, peritoneal primary or fallopian tube cancer.

SECONDARY OBJECTIVES:

I. To determine if the addition of bevacizumab to the second-line and maintenance phase of treatment increases the duration of progression-free survival relative to second-line paclitaxel and carboplatin alone in patients with recurrent platinum sensitive epithelial ovarian cancer, peritoneal primary or fallopian tube cancer.

II. To prospectively determine the incidence of carboplatin and paclitaxel hypersensitivity in these patients undergoing retreatment with both agents as first recurrence therapy.

III. To determine if surgical secondary cytoreduction in addition to adjuvant chemotherapy increases quality of life (QOL) in patients with recurrent platinum-sensitive epithelial ovarian cancer, peritoneal primary or fallopian tube cancer, as measured by the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) trial outcome index and Rand Short Form (SF)-36 physical functioning scale.

IV. To determine if the addition of bevacizumab to the second-line and maintenance phases of treatment increases QOL relative to second-line paclitaxel and carboplatin alone in patients with recurrent platinum-sensitive epithelial ovarian, peritoneal primary or fallopian tube cancer.

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To define molecular and biochemical profiles associated with the duration of progression-free survival in platinum-sensitive recurrent ovarian, peritoneal primary or fallopian tube carcinoma treated with combination chemotherapy with or without bevacizumab followed with or without maintenance bevacizumab therapy in the presence or absence of secondary surgical cytoreduction.

II. To identify molecular determinants that predict sensitivity or resistance to carboplatin and paclitaxel with or without bevacizumab followed with or without maintenance bevacizumab therapy.

III. To bank deoxyribonucleic acid (DNA) from whole blood for research and evaluate the association between single nucleotide polymorphisms (SNPs) and measures of clinical outcome including overall survival, progression-free survival and adverse events.

OUTLINE: Patients are assigned to 1 of 4 treatment groups. Patients who are not candidates for surgical cytoreduction (i.e., those for whom complete cytoreduction in the estimation of the investigator is impossible or a medical infirmity precludes exploration and debulking) are eligible to receive chemotherapy after randomization.

Patients who are eligible for surgery undergo abdominal exploration with cytoreduction. Patients are then randomized to 1 of 4 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours or docetaxel IV over 1 hour and carboplatin IV over 60 minutes on day 1.

ARM II: Patients receive chemotherapy as in Arm I and bevacizumab IV over 30-90 minutes on day 1.

ARM III: Patients receive gemcitabine hydrochloride IV over 60 minutes on days 1 and 8 and carboplatin as in Arm I.

ARM IV: Patients receive gemcitabine hydrochloride IV as in Arm III, bevacizumab IV and carboplatin IV as in Arm II.

In all arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with measurable disease achieving a clinical response (CR) receive 6-8 courses of therapy. Patients with stable disease or partial regression receive a maximum of 8 courses.

Patients without measurable lesions as determined by a computed tomography (CT) scan prior to initiating study treatment continue therapy for 6 courses or, if cancer antigen (CA)-125 normalizes, for 2 courses beyond CA-125 normalization, whichever is greater. Patients in Arm II then receive a maintenance regimen comprising bevacizumab IV over 30-90 minutes. Treatment with bevacizumab alone repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled after August 28, 2011 must be candidates for cytoreductive surgery and consent to have their surgical treatment determined by randomization
* Patients must have histologic diagnosis of epithelial ovarian carcinoma, peritoneal primary or fallopian tube carcinoma, which is now recurrent
* Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's tumor, or adenocarcinoma not otherwise specified (N.O.S.)
* Patients must have had a complete response to front-line platinum-taxane therapy (at least three cycles)
* A complete response to front-line chemotherapy must include: negative physical exam, negative pelvic exam and normalization of CA125, if elevated at baseline; although not required, any radiographic assessment of disease status (e.g. CT, magnetic resonance imaging [MRI], positron emission tomography [PET]/CT, etc) obtained following the completion of primary therapy should be considered negative for disease
* All patients must have also had a treatment-free interval without clinical evidence of progressive disease of at least 6 months from completion of front-line chemotherapy (both platinum and taxane); front-line therapy may have included a biologic agent (i.e. bevacizumab)
* Front-line treatment may include maintenance therapy following complete clinical or pathological response; however, maintenance cytotoxic chemotherapy must be discontinued for a minimum of 6 months prior to documentation of recurrent disease; patients receiving maintenance biological therapy or hormonal therapy are ELIGIBLE provided their recurrence is documented more than 6 months from primary cytotoxic chemotherapy completion (includes maintenance chemotherapy) AND a minimum 4 weeks has elapsed since their last infusion of biological therapy
* Patients must have clinically evident recurrent disease for the purpose of this study
* Measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST]) is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be more than or equal to 20 mm when measured by conventional techniques, MRI or CT, or more than or equal to 10 mm when measured by spiral CT
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3, equivalent to Common Toxicity Criteria for Adverse Events version (v)4.0 (CTCAE) grade 1
* Platelets greater than or equal to 100,000/mm^3 (CTCAE grade 0-1)
* Creatinine (non-isotope dilution mass spectrometry [IDMS]) =< 1.5 x institutional upper limit normal (ULN), CTCAE grade 1
* Total bilirubin =< 1.5 ULN (CTCAE grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) =< 2.5 times the upper limit of normal in the absence of liver metastasis; SGOT/AST < 5.0 times ULN in the presence of liver metastasis
* Alkaline phosphatase =< 2.5 times the upper limit of normal in the absence of liver metastasis; alkaline phosphatase < 5.0 times ULN in the presence of liver metastasis
* This criterion applies only to the patients enrolled before August 29, 2011 and those enrolled after this date electing to receive bevacizumab; patients must have a urine protein-to-creatinine ratio (UPCR) < 1.0 mg/dL
* This eligibility criterion does not apply to patients enrolled after August 28, 2011; patients who are not candidates for surgical cytoreduction are eligible for the chemotherapy randomization; patients are not considered candidates for surgical cytoreduction if complete cytoreduction in the estimation of the investigator is impossible or a medical infirmity precludes exploration and debulking
* Patients must have met the pre-entry requirements as specified
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2

Exclusion Criteria:

* Patients who have received more than one previous regimen of chemotherapy (maintenance is not considered a second regimen)
* Patients receiving concurrent immunotherapy, or radiotherapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded
* Patients whom have already undergone secondary cytoreduction for recurrent disease are excluded
* Patients with a prior histologic diagnosis of borderline, low malignant potential (grade 0) epithelial carcinoma that was surgically resected and who subsequently developed an unrelated, new invasive epithelial ovarian or peritoneal primary cancer are eligible provided that they meet the criteria listed above
* Patients who require parenteral hydration or nutrition and have evidence of partial bowel obstruction or perforation
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor (other than ovarian, fallopian tube, and primary peritoneal) are excluded
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients with uncontrolled infection
* Patients with concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy
* Patients with >= grade 2 peripheral neuropathy
* Patients with a history of allergic reactions to carboplatin and/or paclitaxel or chemically similar compounds; patients with allergic (hypersensitivity) reactions to these chemotherapeutic agents are NOT excluded IF they were successfully retreated following a desensitization program or protocol
* This criterion applies only to the patients enrolled before August 29, 2011 and those enrolled after this date electing to receive bevacizumab; patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients of childbearing potential, not practicing adequate contraception, patients who are pregnant or patients who are nursing are not eligible for this trial; to date, no fetal studies in animal or humans have been performed; the possibility of harm to a fetus is likely; bevacizumab specifically inhibits VEGF, which is responsible for the formation of new blood vessels during development, and antibodies can cross the placenta; therefore, bevacizumab should not be administered to pregnant women; in addition, there are unknown immediate and long-term consequences of chemotherapy administration to these women; in addition, surgical exploration as mandated by randomization during pregnancy may cause imminent mortal consequences; further, it is not known whether bevacizumab is excreted in human milk; because many drugs are excreted in human milk, bevacizumab should not be administered to nursing women; subjects will be apprised of the large potential risk to a developing fetus
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy
* This criterion applies only to the patients enrolled before August 29, 2011 and those enrolled after this date electing to receive bevacizumab; patients with active bleeding or pathologic conditions that carry high risk of bleeding such as a known bleeding disorder, coagulopathy, or tumor involving major vessels
* This criterion applies only to the patients enrolled before August 29, 2011 and those enrolled after this date electing to receive bevacizumab; patients with a history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases or a history of stroke within 5 years of the first date of treatment on this study
* This criterion applies only to the patients enrolled before August 29, 2011 and those enrolled after this date electing to receive bevacizumab; patients with clinically significant cardiovascular disease; this includes:

  * Patients with significant cardiac conduction abnormalities, i.e. PR interval > 0.24 seconds (sec) or 2nd or 3rd degree atrioventricular (AV) block
  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg
  * Myocardial infarction, cardiac arrhythmia or unstable angina < 6 months prior to registration
  * New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Grade II or greater peripheral vascular disease (exception: episodes of ischemia < 24 hours [hrs] in duration, that are managed non-surgically and without permanent deficit)
  * History of cerebrovascular attack (CVA) within six months
* This criterion applies only to the patients enrolled before August 29, 2011 and those enrolled after this date electing to receive bevacizumab; patients who have had a major surgical procedure, open biopsy, dental extractions or other dental surgery/procedure that results in an open wound, or significant traumatic injury within 28 days prior to the first date of treatment on this study, or anticipation of need for major surgical procedure during the course of the study; patients with placement of vascular access device or core biopsy within 7 days prior to the first date of treatment on this study
* Patients undergoing pre-treatment secondary cytoreduction will undergo therapy with bevacizumab on cycle #2
* Patients undergoing pre-treatment surgery for purposes other than cytoreduction may also participate provided they meet eligibility; patients randomized to arms containing bevacizumab must wait a minimum of 28 days since that procedure to begin protocol treatment; patients who undergo an uncomplicated port placement must wait a minimum of 7 days to begin protocol treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2007-12-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2028-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Coleman, Principal Investigator — NRG Oncology
Locations (709):
- United States (680):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - John Muir Medical Center-Concord, Concord, California
  - Sutter Davis Hospital, Davis, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - GenesisCare USA - FGO, Fort Myers, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Abben Cancer Center, Spencer, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Saint Luke's Hospital-Warren Campus, Phillipsburg, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Clinic-Tulsa South, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - Women's Cancer Center of Seattle, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Cancer Institutes of Washington PLLC, Yakima, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
- Japan (16):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Kure Medical Center and Chugoku Cancer Center, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Shizuoka Cancer Center, Shizuoka, Suntou
  - Keio University, Shinjuku-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Shikoku Cancer Center, Matsuyama
  - National Kyushu Cancer Center, Minamiku
  - Jikei University School of Medicine, Minato-ku, Tokyo
  - Kindai University, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - Tottori University, Tottori
- South Korea (13):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Korea
  - Catholic University of Korea-Seoul Saint Mary's Hospital, Seoul, Korea
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Ewha Woman's University, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Coleman RL, Spirtos NM, Enserro D, Herzog TJ, Sabbatini P, Armstrong DK, Kim JW, Park SY, Kim BG, Nam JH, Fujiwara K, Walker JL, Casey AC, Alvarez Secord A, Rubin S, Chan JK, DiSilvestro P, Davidson SA, Cohn DE, Tewari KS, Basen-Engquist K, Huang HQ, Brady MF, Mannel RS. Secondary Surgical Cytoreduction for Recurrent Ovarian Cancer. N Engl J Med. 2019 Nov 14;381(20):1929-1939. doi: 10.1056/NEJMoa1902626. PMID 31722153
- [Derived] Coleman RL, Brady MF, Herzog TJ, Sabbatini P, Armstrong DK, Walker JL, Kim BG, Fujiwara K, Tewari KS, O'Malley DM, Davidson SA, Rubin SC, DiSilvestro P, Basen-Engquist K, Huang H, Chan JK, Spirtos NM, Ashfaq R, Mannel RS. Bevacizumab and paclitaxel-carboplatin chemotherapy and secondary cytoreduction in recurrent, platinum-sensitive ovarian cancer (NRG Oncology/Gynecologic Oncology Group study GOG-0213): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Jun;18(6):779-791. doi: 10.1016/S1470-2045(17)30279-6. Epub 2017 Apr 21. PMID 28438473
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the beginning of the study participants could be randomized to chemotherapy. On August 29, 2011 randomization to chemotherapy ended and participants could only be randomized to surgery.
Groups:
- Arm I (no Surgery; Carboplatin and Paclitaxel): Patients receive paclitaxel IV over 3 hours or docetaxel IV over 1 hour and carboplatin over 30 minutes on day 1. Treatment repeats every 21 days. Patients are not in secondary cytoreductive surgery portion of study.
- Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab): Patients receive chemotherapy as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days. Patients are not in secondary cytoreductive surgery portion of study.
- Arm III (Surgery; Carboplatin and Paclitaxel); Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab): Patients receive paclitaxel IV over 3 hours or docetaxel IV over 1 hour and carboplatin over 30 minutes on day 1. Treatment repeats every 21 days. Patients receive secondary cytoreductive surgery.
- Arm V (no Surgery; Carboplatin and Gemcitabine): Patients receive carboplatin as in arm I. Patients receive gemcitabine. Treatment repeats every 21 days. Patients do not receive secondary cytoreductive surgery.
- Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab): Patients receive carboplatin as in arm I and bevacizumab IV over 30-90 minutes on day 1. Patients receive gemcitabine. Treatment repeats every 21 days. Patients do not receive secondary cytoreductive surgery.
- Arm VII (Surgery; Carboplatin and Gemcitabine): Patients receive carboplatin as in arm I. Patients receive gemcitabine. Treatment repeats every 21 days. Patients receive secondary cytoreductive surgery.
- Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab): Patients receive carboplatin as in arm I and bevacizumab IV over 30-90 minutes on day 1. Patients receive gemcitabine. Treatment repeats every 21 days. Patients receive secondary cytoreductive surgery.
Period: Surgical Assignment
Arm/Group | Arm I (no Surgery; Carboplatin and Paclitaxel) | Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm III (Surgery; Carboplatin and Paclitaxel) | Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm V (no Surgery; Carboplatin and Gemcitabine) | Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab) | Arm VII (Surgery; Carboplatin and Gemcitabine) | Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab)
Started | 316 | 456 | 33 | 165 | 6 | 34 | 5 | 37
Randomized - Yes Surgery | 0 | 0 | 33 | 165 | 0 | 0 | 5 | 37
Randomized - no Surgery | 33 | 172 | 0 | 0 | 6 | 34 | 0 | 0
Not Surgical Candidate | 283 | 284 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Includes participants who followed through with surgical assignment) | 313 | 454 | 31 | 154 | 6 | 34 | 5 | 35
Not Completed | 3 | 2 | 2 | 11 | 0 | 0 | 0 | 2
Period: Chemotherapy Assignment
Arm/Group | Arm I (no Surgery; Carboplatin and Paclitaxel) | Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm III (Surgery; Carboplatin and Paclitaxel) | Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm V (no Surgery; Carboplatin and Gemcitabine) | Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab) | Arm VII (Surgery; Carboplatin and Gemcitabine) | Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab)
Started | 316 | 456 | 33 | 165 | 6 | 34 | 5 | 37
Randomized to Chemo | 310 | 311 | 27 | 26 | 0 | 0 | 0 | 0
Pre-specified Chemo | 6 | 145 | 6 | 139 | 6 | 34 | 5 | 37
Completed | 307 | 433 | 30 | 129 | 6 | 31 | 5 | 34
Not Completed | 9 | 23 | 3 | 36 | 0 | 3 | 0 | 3
Not completed — Never Initiated Chemotherapy | 9 | 9 | 3 | 18 | 0 | 2 | 0 | 2
Not completed — Still On Chemotherapy | 0 | 14 | 0 | 18 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled
Groups:
- Arm I (no Surgery; Carboplatin and Paclitaxel): Patients receive paclitaxel IV over 3 hours or docetaxel IV over 1 hour and carboplatin over 30 minutes on day 1. Treatment repeats every 21 days. Patients are not in secondary cytoreductive surgery portion of study.
  Carboplatin: Given IV
  Docetaxel: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Quality-of-Life Assessment: Ancillary studies
- Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab): Patients receive chemotherapy as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days. Patients are not in secondary cytoreductive surgery portion of study.
  Bevacizumab: Given IV
  Carboplatin: Given IV
  Docetaxel: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Quality-of-Life Assessment: Ancillary studies
- Arm III (Surgery; Carboplatin and Paclitaxel): Patients receive paclitaxel IV over 3 hours or docetaxel IV over 1 hour and carboplatin over 30 minutes on day 1. Treatment repeats every 21 days. Patients receive secondary cytoreductive surgery.
  Carboplatin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Quality-of-Life Assessment: Ancillary studies
- Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab): Patients receive paclitaxel IV over 3 hours or docetaxel IV over 1 hour and carboplatin over 30 minutes on day 1. Treatment repeats every 21 days. Patients receive secondary cytoreductive surgery.
  Bevacizumab: Given IV
  Carboplatin: Given IV
  Docetaxel: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Quality-of-Life Assessment: Ancillary studies
- Arm V (no Surgery; Carboplatin and Gemcitabine): Patients receive carboplatin as in arm I. Patients receive gemcitabine. Treatment repeats every 21 days. Patients do not receive secondary cytoreductive surgery.
  Carboplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
- Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab)): Patients receive carboplatin as in arm I and bevacizumab IV over 30-90 minutes on day 1. Patients receive gemcitabine. Treatment repeats every 21 days. Patients do not receive secondary cytoreductive surgery.
  Bevacizumab: Given IV
  Carboplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
- Arm VII (Surgery; Carboplatin and Gemcitabine): Patients receive carboplatin as in arm I. Patients receive gemcitabine. Treatment repeats every 21 days. Patients receive secondary cytoreductive surgery.
  Carboplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
- Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab)): Patients receive carboplatin as in arm I and bevacizumab IV over 30-90 minutes on day 1. Patients receive gemcitabine. Treatment repeats every 21 days. Patients receive secondary cytoreductive surgery.
  Bevacizumab: Given IV
  Carboplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Arm I (no Surgery; Carboplatin and Paclitaxel) | Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm III (Surgery; Carboplatin and Paclitaxel) | Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm V (no Surgery; Carboplatin and Gemcitabine) | Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab)) | Arm VII (Surgery; Carboplatin and Gemcitabine) | Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab)) | Total
Number analyzed (Participants) | 316 | 456 | 33 | 165 | 6 | 34 | 5 | 37 | 1052
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (10.0) | 59.0 (10.3) | 58.7 (10.0) | 57.1 (10.5) | 72.1 (7.4) | 58.7 (8.2) | 60.7 (9.3) | 61.1 (9.5) | 59.4 (10.2)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 4 | 14 | 0 | 7 | 0 | 0 | 0 | 0 | 25
  40 - 49 years | 40 | 68 | 6 | 37 | 0 | 6 | 1 | 6 | 164
  50 - 59 years | 102 | 170 | 11 | 57 | 1 | 14 | 1 | 9 | 365
  60 - 69 years | 111 | 143 | 10 | 44 | 0 | 12 | 2 | 13 | 335
  70 - 79 years | 52 | 54 | 6 | 19 | 5 | 2 | 1 | 9 | 148
  ≥ 80 years | 7 | 7 | 0 | 1 | 0 | 0 | 0 | 0 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316 | 456 | 33 | 165 | 6 | 34 | 5 | 37 | 1052
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 22 | 0 | 6 | 0 | 0 | 0 | 4 | 46
  Not Hispanic or Latino | 272 | 409 | 30 | 155 | 6 | 34 | 5 | 32 | 943
  Unknown or Not Reported | 30 | 25 | 3 | 4 | 0 | 0 | 0 | 1 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Asian | 39 | 136 | 6 | 101 | 0 | 14 | 1 | 10 | 307
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 15 | 17 | 1 | 4 | 1 | 3 | 1 | 2 | 44
  White | 255 | 294 | 26 | 57 | 5 | 17 | 3 | 25 | 682
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 20 | 108 | 4 | 90 | 0 | 11 | 0 | 9 | 242
  United States | 284 | 324 | 29 | 67 | 6 | 23 | 5 | 28 | 766
  Japan | 12 | 24 | 0 | 7 | 0 | 0 | 0 | 0 | 43
  Russia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Histology [Count of Participants; unit: Participants]
  Serous | 252 | 383 | 30 | 142 | 5 | 30 | 4 | 35 | 881
  Endometrioid | 25 | 24 | 0 | 9 | 1 | 2 | 0 | 2 | 63
  Clear Cell | 13 | 14 | 1 | 5 | 0 | 0 | 0 | 0 | 33
  Mucinous | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Other | 24 | 33 | 2 | 9 | 0 | 2 | 1 | 0 | 71

OUTCOME MEASURES:

1. Primary Outcome: To Determine if Surgical Secondary Cytoreduction in Addition to Adjuvant Chemotherapy Increases the Duration of Overall Survival in Patients With Recurrent Platinum Sensitive Epithelial Ovarian Cancer, Peritoneal Primary or Fallopian Tube Cancer
Description: The treatment regimens will be compared with a logrank procedure which includes all of the patients categorized by their randomly assigned treatment. The logrank test will be stratified by the secondary surgical debulking status (randomized to undergo cytoreduction, vs randomized to not undergo secondary cytoreduction vs not a candidate or did not consent to secondary surgical cytoreduction) and the duration of treatment free-interval prior to enrolling onto this study (6-12 months vs > 12 months). The median duration of follow-up is calculated by the reverse Kaplan-Meier method.
Time Frame: The time frame is 82.5 months (median duration of follow-up)
Population: All patients who were eligible for the surgery analysis (data were combined and analyzed according to randomized surgical assignment, regardless of chemotherapy regimen, as pre-specified in the study protocol)
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- No Cytoreductive Surgery: All patients enrolled in the study who did not receive cytoreductive surgery and included in the surgery analysis
- Cytoreductive Surgery: All patients enrolled in the study who received secondary cytoreductive surgery and were included in the surgery analysis
Arm/Group | No Cytoreductive Surgery | Cytoreductive Surgery
Number analyzed (Participants) | 245 | 240
Months | 64.7 [54.5 to 73.9] | 50.6 [44.2 to 59.7]

2. Primary Outcome: To Determine if the Addition of Bevacizumab Increases the Duration of Overall Survival Relative to Second-line Paclitaxel and Carboplatin Alone in Patients With Recurrent Platinum Sensitive Epithelial Ovarian, Peritoneal Primary or Fallopian Tube Cancer
Description: as for outcome 1
Time Frame: The time frame is 82.5 months (median duration of follow-up).
Population: All patients who were enrolled between December 10, 2007 and August 26, 2011 and received paclitaxel and carboplatin (with or without bevacizumab) (data were combined and analyzed according to randomized chemotherapy regimen, regardless of surgical assignment, as pre-specified in the study protocol).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Paclitaxel and Carboplatin Chemotherapy: All patients who received paclitaxel and carboplatin chemotherapy and were included in the chemotherapy analysis
- Paclitaxel and Carboplatin Chemotherapy With Bevacizumab: All patients who received paclitaxel and carboplatin chemotherapy with bevacizumab followed by bevacizumab maintenance therapy and were included in the chemotherapy analysis
Arm/Group | Paclitaxel and Carboplatin Chemotherapy | Paclitaxel and Carboplatin Chemotherapy With Bevacizumab
Number analyzed (Participants) | 337 | 337
Months | 37.3 [32.6 to 39.7] | 42.2 [37.7 to 46.2]

3. Secondary Outcome: Progression-free Survival (Chemotherapy Analysis)
Description: Progression-free survival was defined as the time from randomization to cancer progression as shown on radiography, according to the RECIST version 1.0 criteria, an increase in the CA125 level according to Gynecologic Cancer InterGroup (GCIG) criteria, global deterioration of health, or death from any cause.
Time Frame: Radiographic assessment of disease was conducted during chemotherapy and then every 6 months during the maintenance / surveillance phase
Population: All patients who were enrolled and eligible for the chemotherapy analysis (data were combined and analyzed according to randomized chemotherapy regimen, regardless of surgical assignment, as pre-specified in the study protocol).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel and Carboplatin Chemotherapy | Paclitaxel and Carboplatin Chemotherapy With Bevacizumab
Number analyzed (Participants) | 337 | 337
Months | 10.4 [9.7 to 11.0] | 13.8 [13.0 to 14.7]

4. Secondary Outcome: Progression Free Survival (Surgery Analysis)
Description: as for outcome 3
Time Frame: Radiographic assessment of disease (in patients with measurable and non-measurable disease) was conducted Every three months for two years and then every 6 months after completion of chemotherapy during the maintenance/surveillance phase.
Population: All randomized patients who were eligible for the surgery analysis (data were combined and analyzed according to randomized surgical assignment, regardless of chemotherapy regimen, as pre-specified in the study protocol).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | No Cytoreductive Surgery | Cytoreductive Surgery
Number analyzed (Participants) | 245 | 240
Months | 16.2 [14.2 to 19.6] | 18.9 [16.8 to 21.0]

5. Secondary Outcome: Summary of Adverse Events (CTCAE Version 4.0)
Description: Number of treated patients with at least one adverse event reported (assessed by Common Terminology Criteria for Adverse Events (version 4.0))
Time Frame: During treatment period and up to 100 days after stopping the study treatment, a median duration of 82.5 months
Population: Eligible and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (no Surgery; Carboplatin and Paclitaxel) | Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm III (Surgery; Carboplatin and Paclitaxel) | Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm V (no Surgery; Carboplatin and Gemcitabine) | Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab)) | Arm VII (Surgery; Carboplatin and Gemcitabine) | Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab))
Number analyzed (Participants) | 316 | 456 | 33 | 165 | 6 | 34 | 5 | 37
Participants | 304 | 376 | 29 | 77 | 3 | 9 | 3 | 9

6. Secondary Outcome: Patient Reported Quality of Life (Chemotherapy Analysis)
Description: Patient reported quality of life was measured with the Treatment Outcome Index (TOI) of the Functional Assessment of Cancer Therapy for ovarian cancer (FACT-O TOI). The FACT-O TOI is a scale for assessing general QOL of ovarian cancer patients. It consists of three subscales: Physical Well Being (7 items), Functional Well Being (7 items), and Ovarian Cancer subscale (11 items). Each item in the FACT-O TOI was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). The FACT-O TOI score ranges 0-100 with a large score suggests better QOL.
Time Frame: 1. Prior to cycle 1 (baseline), 2. Prior to cycle 3 (6 weeks post cycle 1), 3. Prior to cycle 6 (15 weeks post cycle 1), 4. 6 months post cycle 1, 5. 12 months post cycle 1.
Population: Provided baseline and at least one follow-up assessment (data were combined and analyzed according to randomized chemotherapy regimen, regardless of surgical assignment, as pre-specified in the study protocol).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Paclitaxel and Carboplatin Chemotherapy | Paclitaxel and Carboplatin Chemotherapy With Bevacizumab
Number analyzed (Participants) | 298 | 302
score on a scale
  Prior to cycle 1 (baseline) | 75.8 (0.8) | 75.3 (0.9)
  Prior to cycle 3 | 74.2 (1.0) | 73.4 (0.9)
  Prior to cycle 6 | 73.3 (1.0) | 72.3 (1.0)
  6 months post cycle 1 | 77.1 (1.0) | 77.2 (1.0)
  12 months post cycle 1 | 77.0 (1.1) | 77.8 (1.0)

7. Secondary Outcome: Patient Reported Physical Function (Chemotherapy Analysis)
Description: Patient reported physical functioning was measured with physical functioning subscale of the RAND SF-36. The Physical Functioning Subscale consists of 10 items concerning activities of daily living: walking, climbing stairs, bathing, dressing, and performance of physical activities. Each item is rated on a three-point scale of limitation of activity due to the patients' health from 1=limited a lot to 3=not limited. The total PF score is the summation of item scores and then rescaled to 0-100. A larger score suggests better physical functioning.
Time Frame: as for outcome 6
Population: Provided baseline and at least one follow-up assessments (data were combined and analyzed according to randomized chemotherapy regimen, regardless of surgical assignment, as pre-specified in the study protocol).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Paclitaxel and Carboplatin Chemotherapy | Paclitaxel and Carboplatin Chemotherapy With Bevacizumab
Number analyzed (Participants) | 298 | 302
score on a scale
  Prior to cycle 1 (baseline) | 71.5 (1.6) | 69.4 (1.7)
  Prior to cycle 3 | 73.2 (2.1) | 69.8 (2.1)
  Prior to cycle 6 | 71.5 (2.2) | 64.6 (2.2)
  6 months post cycle 1 | 71.6 (2.2) | 70.2 (2.1)
  12 months post cycle 1 | 71.8 (2.2) | 70.7 (2.2)

8. Secondary Outcome: Patient Reported Quality of Life (Surgery Analysis)
Description: as for outcome 6
Time Frame: 1. Prior to surgery, 2. 6 weeks post-surgery, 3. 15 weeks post-surgery, 4. 6 months post-surgery, 5. 12 months post-surgery.
Population: Provided baseline and at least one follow-up assessment (data were combined and analyzed according to randomized surgical assignment, regardless of chemotherapy regimen, as pre-specified in the study protocol).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | No Cytoreductive Surgery | Cytoreductive Surgery
Number analyzed (Participants) | 215 | 206
score on a scale
  Prior to surgery | 74.5 (1.0) | 74.2 (1.0)
  6 weeks post-surgery | 69.3 (1.3) | 68.4 (1.3)
  15 weeks post-surgery | 68.7 (1.3) | 68.8 (1.3)
  6 months post-surgery | 72.6 (1.3) | 73.5 (1.3)
  12 months post-surgery | 74.0 (1.4) | 75.6 (1.3)

9. Secondary Outcome: Patient Reported Physical Functioning (Surgery Analysis)
Description: Patient reported physical functioning was measured with physical functioning subscale of the RAND SF-36. The Physical Functioning subscale consists of 10 items concerning activities of daily living: walking, climbing stairs, bathing, dressing, and performance of physical activities. Each item is rated on a three-point scale of limitation of activity due to the patients' health from 1=limited a lot to 3=not limited. The total PF score is the summation of item scores and then rescaled to 0-100. A larger score suggests better physical functioning. This measure was completed by US patients only.
Time Frame: 1. Prior to surgery (baseline), 2. 6 weeks post-surgery, 3. 15 weeks post-surgery 4. 6 months post-surgery, 5. 12 months post-surgery
Population: US patients who provided baseline and ≥ 1 follow-up assessments (data were combined and analyzed according to randomized surgical assignment, regardless of chemotherapy regimen, as pre-specified in the study protocol).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | No Cytoreductive Surgery | Cytoreductive Surgery
Number analyzed (Participants) | 104 | 113
score on a scale
  Prior to surgery (baseline) | 73.4 (2.3) | 71.7 (2.3)
  6 weeks post-surgery | 73.2 (2.1) | 69.8 (2.1)
  15 weeks post-surgery | 71.5 (2.2) | 64.6 (2.2)
  6 months post-surgery | 71.6 (2.2) | 70.2 (2.1)
  12 months post-surgery | 71.8 (2.2) | 70.7 (2.2)

ADVERSE EVENTS:
Time Frame: During treatment period and up to 100 days after stopping the study treatment, a median duration of 82.5 months.
Description: Eligible and treated participants were affected if they experienced grade 1 - 5 adverse event. Adverse events were not collected in a manner that allow them to be attributed to an intervention (i.e. surgery or chemotherapy).
Arm/Group | Arm I (no Surgery; Carboplatin and Paclitaxel) | Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm III (Surgery; Carboplatin and Paclitaxel) | Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab) | Arm V (no Surgery; Carboplatin and Gemcitabine) | Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab) | Arm VII (Surgery; Carboplatin and Gemcitabine) | Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 253/316 | 299/456 | 28/33 | 56/165 | 4/6 | 14/34 | 4/5 | 21/37
Serious Adverse Events (participants affected / at risk) | 37/316 | 104/456 | 1/33 | 24/165 | 0/6 | 1/34 | 2/5 | 2/37
Other Adverse Events (participants affected / at risk) | 304/316 | 376/456 | 29/33 | 77/165 | 3/6 | 9/34 | 3/5 | 9/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (no Surgery; Carboplatin and Paclitaxel) (N=316) | Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab) (N=456) | Arm III (Surgery; Carboplatin and Paclitaxel) (N=33) | Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab) (N=165) | Arm V (no Surgery; Carboplatin and Gemcitabine) (N=6) | Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab) (N=34) | Arm VII (Surgery; Carboplatin and Gemcitabine) (N=5) | Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab) (N=37)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1 | 8 | 0 | 2 | 0 | 0 | 1 | 0
Myelodysplasia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophils (Blood and lymphatic system disorders) | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Platelets (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytes (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Cardiac disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardipulmonary Arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death No Ctcae Term - Disease Progression Nos (General disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Death No Ctcae Term - Death Nos (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death No Ctcae Term - Sudden Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Perforation, Gi - Colon (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dental: Periodontal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction, Gi - Colon (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Perforation, Gi - Cecum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ulcer,gi - Stomach (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 6 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Rectum (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Stomach (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Cns (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Foreign Body (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Soft Tissue Nos (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Febrile Neutropenia (Infections and infestations) | 7 | 14 | 0 | 3 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection - Other (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inf Unknown Anc: Liver (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Foreign Body (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Foreign Body (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Eye Nos (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholesterol,serum High (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alt (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Weakness - Right-Sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neurology - Other (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mood Alteration - Depression (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cns Ischemia (Nervous system disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Confusion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy-Sensory (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy-Motor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blurred Vision (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain - Other (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Chest /Thorax Nos (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Head/Headache (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Back (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain: Abdominal Pain Nos (General disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular - Other (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 4 | 6 | 0 | 1 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (no Surgery; Carboplatin and Paclitaxel) (N=316) | Arm II (no Surgery; Carboplatin, Paclitaxel and Bevacizumab) (N=456) | Arm III (Surgery; Carboplatin and Paclitaxel) (N=33) | Arm IV (Surgery; Carboplatin, Paclitaxel and Bevacizumab) (N=165) | Arm V (no Surgery; Carboplatin and Gemcitabine) (N=6) | Arm VI (no Surgery; Carboplatin, Gemcitabine and Bevacizumab) (N=34) | Arm VII (Surgery; Carboplatin and Gemcitabine) (N=5) | Arm VIII (Surgery; Carboplatin, Gemcitabine and Bevacizumab) (N=37)
Allergy/Immunology - Other (Immune system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Allergic Reaction/Hypersensitivity (Immune system disorders) | 76 | 86 | 6 | 16 | 1 | 0 | 1 | 3
Vasculitis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Immune system disorders) | 13 | 62 | 1 | 8 | 0 | 0 | 0 | 1
Autoimmune Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Middle Ear (Ear and labyrinth disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 5 | 12 | 1 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 15 | 23 | 1 | 2 | 1 | 0 | 1 | 0
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophils (Blood and lymphatic system disorders) | 282 | 363 | 28 | 72 | 3 | 7 | 3 | 8
Platelets (Blood and lymphatic system disorders) | 173 | 264 | 22 | 52 | 3 | 7 | 3 | 8
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytes (Blood and lymphatic system disorders) | 276 | 350 | 28 | 67 | 3 | 9 | 3 | 9
Lymphopenia (Blood and lymphatic system disorders) | 21 | 31 | 1 | 2 | 0 | 0 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 279 | 316 | 29 | 67 | 3 | 9 | 3 | 9
Prolonged Qtc Interval (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 12 | 19 | 1 | 4 | 1 | 0 | 1 | 0
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 5 | 15 | 1 | 1 | 0 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular Arrhythmia - Pvcs (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Arrhythmia - Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Cardiac disorders) | 10 | 147 | 0 | 22 | 0 | 1 | 1 | 5
Restrictive Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac General - Other (Cardiac disorders) | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Cardiac Troponin I (Ctni) (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 3 | 12 | 0 | 1 | 0 | 0 | 0 | 0
Cardipulmonary Arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inr (Vascular disorders) | 1 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Dic (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic Microangiopathy (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ptt (Vascular disorders) | 1 | 7 | 1 | 0 | 0 | 0 | 0 | 0
Constitutional Symptoms - Other (General disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Sweating (General disorders) | 10 | 8 | 2 | 2 | 0 | 0 | 0 | 0
Weight Gain (General disorders) | 18 | 27 | 1 | 6 | 0 | 0 | 0 | 1
Fever (General disorders) | 31 | 45 | 1 | 13 | 0 | 0 | 0 | 0
Weight Loss (General disorders) | 12 | 54 | 1 | 6 | 0 | 0 | 1 | 0
Rigors/Chills (General disorders) | 7 | 14 | 1 | 3 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 245 | 297 | 25 | 48 | 2 | 5 | 3 | 5
Insomnia (General disorders) | 47 | 67 | 4 | 13 | 0 | 1 | 0 | 3
Nail Changes (Skin and subcutaneous tissue disorders) | 9 | 39 | 0 | 1 | 0 | 1 | 0 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 3 | 9 | 0 | 2 | 0 | 0 | 0 | 0
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 245 | 289 | 21 | 47 | 2 | 3 | 1 | 2
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 0 | 8 | 2 | 2 | 0 | 0 | 1 | 1
Bruising (Skin and subcutaneous tissue disorders) | 11 | 15 | 0 | 1 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 9 | 0 | 2 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 49 | 87 | 4 | 10 | 0 | 3 | 1 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 5 | 25 | 0 | 3 | 0 | 1 | 0 | 1
Decubitus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 46 | 2 | 10 | 0 | 0 | 0 | 1
Burn (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 23 | 0 | 1 | 0 | 1 | 0 | 0
Flushing (Skin and subcutaneous tissue disorders) | 11 | 21 | 1 | 3 | 0 | 0 | 0 | 0
Hand-Foot (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 3 | 0 | 0 | 0 | 0
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 10 | 23 | 0 | 3 | 0 | 0 | 0 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 10 | 0 | 1 | 0 | 0 | 0 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 9 | 0 | 1 | 0 | 0 | 0 | 1
Hot Flashes (Endocrine disorders) | 27 | 45 | 5 | 8 | 0 | 2 | 0 | 1
Diabetes (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adh Secrection Abnormality (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Endocrine - Other (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Salivary Gland Changes (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 5 | 11 | 0 | 0 | 0 | 0 | 0 | 1
Ulcer,gi - Esophagus (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Perforation, Gi - Colon (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental: Periodontal (Gastrointestinal disorders) | 0 | 10 | 0 | 1 | 0 | 0 | 0 | 1
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fistula, Gi - Rectum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 4 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Perforation, Gi - Cecum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 22 | 0 | 1 | 0 | 0 | 0 | 0
Heartburn (Gastrointestinal disorders) | 28 | 51 | 3 | 8 | 0 | 0 | 0 | 0
Mucositis (Functional/Sympt) - Esophagus (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ulcer,gi - Stomach (Gastrointestinal disorders) | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0
Dental: Teeth (Gastrointestinal disorders) | 0 | 7 | 0 | 1 | 0 | 0 | 0 | 0
Mucositis (Functional/Sympt) - Trachea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Leak, Gi - Rectum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 6 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Distention (Gastrointestinal disorders) | 18 | 27 | 3 | 6 | 0 | 0 | 0 | 0
Taste Alteration (Gastrointestinal disorders) | 36 | 46 | 3 | 10 | 0 | 0 | 0 | 1
Incontinence, Anal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 6 | 17 | 0 | 1 | 0 | 0 | 0 | 1
Mucositis (Functional/Sympt) - Stomach (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis (Functional/Sympt) - Rectum (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 32 | 69 | 2 | 8 | 0 | 1 | 0 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Fistula, Gi - Oral Cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 23 | 67 | 0 | 14 | 0 | 4 | 1 | 0
Mucositis (Clinical Exam) - Larynx (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 75 | 125 | 7 | 16 | 0 | 0 | 1 | 4
Anorexia (Gastrointestinal disorders) | 78 | 129 | 10 | 19 | 0 | 3 | 1 | 1
Dehydration (Gastrointestinal disorders) | 12 | 20 | 1 | 5 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 167 | 193 | 20 | 39 | 2 | 2 | 1 | 3
Stricture, Gi - Stomach (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 182 | 223 | 19 | 42 | 1 | 3 | 1 | 6
Gastrointestinal - Other (Gastrointestinal disorders) | 3 | 10 | 1 | 1 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 98 | 148 | 11 | 30 | 0 | 3 | 0 | 4
Ulcer,gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucositis (Clinical Exam) - Pharynx (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gu - Vagina (Vascular disorders) | 8 | 9 | 1 | 1 | 0 | 0 | 0 | 0
Hemorrhage, Gu - Urethra (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage/Pulmonary - Lung (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Rectum (Vascular disorders) | 6 | 19 | 0 | 1 | 0 | 0 | 0 | 0
Hemorrhage/Pulmonary - Respiratory Tract Nos (Vascular disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Hemorrhage, Gi - Stoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Varices (Rectal) (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 8 | 116 | 0 | 13 | 0 | 3 | 0 | 0
Hematoma (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Anus (Vascular disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gu - Ureter (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Lower Gi Nos (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 2 | 17 | 0 | 3 | 0 | 1 | 0 | 0
Hemorrhage, Gu - Bladder (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Stomach (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage, Gi - Colon (Vascular disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Vascular disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 | 3 | 0 | 3 | 0 | 0 | 0 | 0
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver Dysfunction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Middle Ear (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 10 | 20 | 1 | 1 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Nose (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Larynx (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Eye Nos (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Meninges (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Brain (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Soft Tissue Nos (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Joint (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Otitis Media Nos (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 6 | 7 | 1 | 1 | 1 | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Febrile Neutropenia (Infections and infestations) | 2 | 9 | 0 | 2 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Lip/Perioral (Infections and infestations) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Nose (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Sinus (Infections and infestations) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 0 | 7 | 0 | 1 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 19 | 25 | 3 | 2 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Ungual (Nails) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Stomach (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection - Other (Infections and infestations) | 7 | 14 | 1 | 2 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Opportunisitic Inf Assoc. W/Gr 2 Lymphopenia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 1 | 4 | 1 | 2 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Conjunctiva (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Appendix (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 5 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Pharynx (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Bronchus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Eye Nos (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Soft Tissue Nos (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 6 | 10 | 0 | 2 | 0 | 0 | 0 | 0
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inf Unknown Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Foreign Body (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Dental-Tooth (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Abdomen Nos (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Inf Unknown Anc: Middle Ear (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Vulva (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Vagina (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 4 | 6 | 0 | 4 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Anal/Perianal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Sinus (Infections and infestations) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Pharynx (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Nose (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Bronchus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Joint (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 3 | 8 | 1 | 0 | 0 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: External Ear (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphedema-Related Fibrosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphatics - Other (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Edema: Limb (Blood and lymphatic system disorders) | 40 | 44 | 3 | 8 | 1 | 1 | 0 | 3
Edema: Head And Neck (Blood and lymphatic system disorders) | 1 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Ast (Metabolism and nutrition disorders) | 30 | 62 | 2 | 6 | 0 | 2 | 1 | 3
Gfr (Metabolism and nutrition disorders) | 2 | 7 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 10 | 14 | 0 | 1 | 0 | 0 | 0 | 0
Cholesterol,serum High (Metabolism and nutrition disorders) | 2 | 17 | 0 | 2 | 0 | 0 | 1 | 0
Proteinuria (Metabolism and nutrition disorders) | 3 | 70 | 0 | 17 | 0 | 0 | 0 | 0
Creatinine (Metabolism and nutrition disorders) | 17 | 52 | 1 | 5 | 0 | 2 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 | 43 | 1 | 4 | 0 | 3 | 1 | 0
Ggt (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Alt (Metabolism and nutrition disorders) | 27 | 41 | 1 | 5 | 0 | 0 | 2 | 3
Alkaline Phosphatase (Metabolism and nutrition disorders) | 22 | 35 | 2 | 1 | 0 | 1 | 1 | 3
Bilirubin (Metabolism and nutrition disorders) | 3 | 12 | 1 | 0 | 0 | 0 | 0 | 0
Lipase (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 13 | 1 | 2 | 0 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 13 | 22 | 3 | 3 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 19 | 60 | 1 | 2 | 0 | 1 | 1 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 11 | 0 | 2 | 0 | 0 | 1 | 0
Cpk (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 3 | 7 | 0 | 1 | 0 | 0 | 0 | 0
Amylase (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 5 | 5 | 1 | 2 | 0 | 1 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 16 | 48 | 1 | 6 | 0 | 2 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 10 | 26 | 0 | 8 | 0 | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 74 | 111 | 5 | 10 | 1 | 3 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 33 | 48 | 3 | 7 | 0 | 2 | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 7 | 21 | 1 | 3 | 0 | 2 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 6 | 20 | 0 | 5 | 0 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 51 | 104 | 8 | 13 | 0 | 1 | 1 | 1
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1 | 11 | 1 | 1 | 0 | 2 | 0 | 0
Soft Tissue Necrosis - Abdomen (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint-Function (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 3 | 0 | 0 | 0 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Extremity-Upper (Function) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait/Walking (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Spine Rom (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 20 | 1 | 3 | 0 | 0 | 0 | 0
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 15 | 32 | 4 | 6 | 0 | 2 | 0 | 1
Muscle Weakness - Right-Sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Weakness - Left-Sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 8 | 15 | 4 | 2 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 3 | 8 | 1 | 1 | 0 | 0 | 0 | 0
Involuntary Movement (Nervous system disorders) | 5 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Neurology - Other (Nervous system disorders) | 1 | 5 | 0 | 0 | 1 | 0 | 0 | 0
Mental Status (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Mood Alteration - Depression (Nervous system disorders) | 42 | 51 | 5 | 12 | 1 | 1 | 0 | 1
Mood Alteration - Anxiety (Nervous system disorders) | 39 | 57 | 3 | 13 | 0 | 0 | 0 | 1
Mood Alteration - Agitation (Nervous system disorders) | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Speech Impairment (Nervous system disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Cognitive Disturbance (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cns Ischemia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Confusion (Nervous system disorders) | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 7 | 16 | 0 | 3 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 24 | 51 | 4 | 8 | 1 | 2 | 0 | 0
Neuropathy,cranial - Cn Xii Motor-Tongue (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy,cranial - Cn Viii Hearing/Balance (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy,cranial - Cn Vii Motor-Face (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy,cranial - Cn Iii Pupil (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy,cranial - Cn I Smell (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy-Sensory (Nervous system disorders) | 237 | 272 | 18 | 55 | 3 | 4 | 1 | 5
Neuropathy-Motor (Nervous system disorders) | 15 | 14 | 2 | 5 | 1 | 0 | 0 | 0
Ocular/Visual - Other (Eye disorders) | 6 | 11 | 1 | 2 | 1 | 1 | 0 | 0
Scleral Necrosis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Watery Eye (Eye disorders) | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 1 | 5 | 1 | 0 | 0 | 0 | 0 | 0
Ocular Surface Disease (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flashing Lights/Floaters (Eye disorders) | 6 | 19 | 0 | 3 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Blurred Vision (Eye disorders) | 36 | 55 | 2 | 4 | 0 | 1 | 0 | 1
Eyelid Dysfunction (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pain - Other (General disorders) | 6 | 22 | 2 | 3 | 1 | 0 | 0 | 0
Pain: Urethra (General disorders) | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0
Pain: Perineum (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Pelvis (General disorders) | 10 | 11 | 2 | 4 | 0 | 0 | 0 | 0
Pain: Breast (General disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Vagina (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain: Chest /Thorax Nos (General disorders) | 6 | 23 | 1 | 5 | 0 | 0 | 0 | 1
Pain: Chest Wall (General disorders) | 10 | 17 | 1 | 2 | 0 | 0 | 0 | 0
Pain: Throat/Pharynx/Larynx (General disorders) | 9 | 31 | 1 | 4 | 0 | 1 | 0 | 1
Pain: Pleura (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Larynx (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Eye (General disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Head/Headache (General disorders) | 59 | 142 | 7 | 19 | 2 | 4 | 1 | 2
Pain: Neck (General disorders) | 1 | 33 | 0 | 2 | 0 | 0 | 0 | 1
Pain: Extremity-Limb (General disorders) | 41 | 97 | 7 | 13 | 0 | 1 | 0 | 1
Pain: Buttock (General disorders) | 1 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Pain: Back (General disorders) | 35 | 65 | 3 | 13 | 0 | 0 | 1 | 2
Pain: Joint (General disorders) | 99 | 166 | 4 | 28 | 1 | 2 | 0 | 3
Pain: Bone (General disorders) | 19 | 33 | 3 | 8 | 0 | 0 | 0 | 0
Pain: Kidney (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Bladder (General disorders) | 1 | 4 | 2 | 2 | 0 | 0 | 0 | 0
Pain: Pain Nos (General disorders) | 4 | 8 | 0 | 7 | 0 | 0 | 0 | 0
Pain: Stomach (General disorders) | 3 | 9 | 1 | 2 | 0 | 0 | 0 | 0
Pain: Rectum (General disorders) | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Oral Cavity (General disorders) | 2 | 13 | 1 | 4 | 0 | 0 | 0 | 0
Pain: Esophagus (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Dental/Teeth/Peridontal (General disorders) | 0 | 9 | 0 | 1 | 0 | 0 | 0 | 2
Pain: Abdominal Pain Nos (General disorders) | 84 | 127 | 16 | 36 | 2 | 2 | 1 | 4
Pain: Scalp (General disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Oral - Gums (General disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Skin (General disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Pain: Lip (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain: Middle Ear (General disorders) | 5 | 8 | 1 | 1 | 0 | 0 | 0 | 1
Pain: External Ear (General disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Cardiac/ Heart (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Pain: Face (General disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Tumor (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain: Muscle (General disorders) | 55 | 107 | 4 | 23 | 0 | 0 | 0 | 1
Pain: Anus (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain: Neuralgia (General disorders) | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Pain: Sinus (General disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Airway Obstruction - Larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Airway Obstruction - Bronchus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 8 | 50 | 1 | 7 | 1 | 1 | 0 | 2
Edema, Larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 6 | 55 | 0 | 8 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 110 | 5 | 14 | 1 | 2 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 80 | 110 | 4 | 15 | 2 | 1 | 1 | 2
Renal/Genitourinary - Other (Renal and urinary disorders) | 2 | 10 | 1 | 0 | 1 | 0 | 0 | 0
Cystitis (Renal and urinary disorders) | 0 | 10 | 0 | 3 | 0 | 0 | 0 | 0
Urinary Color Change (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 6 | 0 | 1 | 0 | 0 | 0 | 0
Obstruction, Gu - Urethra (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incontinence, Urinary (Renal and urinary disorders) | 16 | 20 | 1 | 3 | 0 | 1 | 0 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 25 | 35 | 3 | 4 | 1 | 1 | 1 | 0
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Libido (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 4 | 7 | 0 | 3 | 0 | 0 | 0 | 0
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginitis (Reproductive system and breast disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 4 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine Release Syndrome (General disorders) | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Flu-Like Syndrome (General disorders) | 1 | 17 | 0 | 4 | 0 | 0 | 0 | 0
Vascular - Other (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Visceral Arterial Ischemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vein Injury - Extremity-Lower (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Artery Injury - Other Nos (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 0 | 11 | 0 | 2 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 5 | 0 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT00565851/Prot_SAP_000.pdf